CLINICAL TRIAL: NCT06603103
Title: Prospective Randomized Study Comparing the SpheriKA® (MEDACTA) and Origin® (SYMBIOS) Prostheses During Total Knee Replacement Using the Kinematic Alignment Technique
Acronym: KAOR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique du Sport, Bordeaux Mérignac (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-21-SBM
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Knee Osteoarthritis
Keywords: Total knee arthroplasty; kinematic alignment; joint perception; biomechanics
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- total knee arthroplasty with kinematic alignment and SPHERIKA prosthesis (Experimental)
  Interventions: Procedure: SPHERIKA prosthesis
- total knee arthroplasty with kinematic alignment and ORIGIN prosthesis (Experimental)
  Interventions: Procedure: ORIGIN prosthesis

INTERVENTIONS:
Procedure: SPHERIKA prosthesis — total knee arthroplasty with kinematic alignement with SPHERIKA prosthesis
  Arms: total knee arthroplasty with kinematic alignment and SPHERIKA prosthesis
Procedure: ORIGIN prosthesis — total knee arthroplasty with kinematic alignement with ORIGIN prosthesis
  Arms: total knee arthroplasty with kinematic alignment and ORIGIN prosthesis

SUMMARY:
The traditional technique for implanting a total knee prosthesis, known as mechanical alignment, does not aim to preserve the original anatomy and laxity of the knee. Instead, the implants are "systematically" aligned to create a non-naturally straight lower limb. Respectively 20% and 50% of patients with a mechanically aligned total knee prosthesis are dissatisfied with the result, and complain of residual symptoms. A newer, more physiological technique for implanting a total knee prosthesis, known as kinematic alignment, aims to recreate the unique native anatomy and laxity of each patient's knee. The kinematic alignment technique has been shown to reduce the risk of residual symptoms and thus improve the patient's experience of his or her prosthetic knee. As a result of the emergence of the kinematic alignment technique, two manufacturers have developed total knee prosthesis implants specifically for this new insertion technique. A "made-to-measure" total knee prosthesis (ORIGIN® - Symbios, Yverdon-les-Bains, Switzerland) was developed with the aim of reproducing the unique contour of each implanted knee. Another manufacturer opted to develop a generic total knee prosthesis implant (SPHERIKA® - Medacta, Castel San Pietro, Switzerland), but with a design optimized for the kinematic alignment technique. These two models of total knee prosthesis each offer advantages and limitations that need to be assessed. The main aim of this study is therefore to compare the joint perception of these 2 prostheses. It will also look at the clinical and imaging results, the biomechanics of the prosthetic knee during gait, and the muscular strength of knee extension, obtained for these 2 total knee prostheses.

ELIGIBILITY:
Inclusion Criteria:

* Patient with indication for initial total knee replacement
* Patient affiliated to a social security scheme
* Patient informed of the study and formally included (informed consent signed) before the first research examination.

Exclusion Criteria:

* Patient with complex osteoarthritis (e.g. bone loss, history of patellar instability)
* Patient with contralateral knee prosthesis
* Patient with symptomatic osteoarthritis (stiffness and/or pain) of a hip or contralateral knee
* Patient with another condition (acquired pathology) of the lower limbs and/or nervous system that may significantly affect gait quality
* Patient deprived of liberty by judicial or administrative decision,
* Patient of legal age under legal protection or unable to express consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-10-03 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Evolution of "forgotten joint score" | 2 months before surgery ; 45 days after surgery ; 1 year after surgery ; 2 years after surgery
  This score consists in 12 questions with a Likert scale from 0 to 5. A high score indicates a high degree of forgetfulness of the prosthesis on the part of the patient.

SECONDARY OUTCOMES:
Frontal alignment of the lower limb | 2 months before surgery ; 45 days after surgery ; 1 year after surgery ; 2 years after surgery
Walking ability | 2 years after surgery
  Evaluation of walking ability : walking speed, cadence, stride length, stride duration
Evaluation of muscular strength | 2 years after surgery
  Measure of :
  * Maximum force developed (N)
  * Explosivity (time required to develop maximum force, N/s)
  * Power (cumulative force developed during the entire acquisition period, W)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique du Sport, Mérignac, France

IPD SHARING:
Plan to Share IPD: No